CLINICAL TRIAL: NCT02744248
Title: A Phase I Study to Determine the MTD and to Evaluate Pharmacokinetic, Safety/Tolerability, and Efficacy Profiles of IOP Injection for MRI Contrast Agent in Healthy Subjects
Brief Title: Phase I , MTD, Pharmacokinetic, Safety/Tolerability, Efficacy of IOP Injection for MRI in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MegaPro Biomedical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: CEECTTA20100721; IOP-CT-001 (Other: MPB)
Record Dates: First submitted 2016-03-24; First posted 2016-04-20 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Magnetic Resonance Imaging
Keywords: Magnetic Resonance Imaging (MRI)
MeSH Terms: interventions — Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IOP Injection (Active Comparator): Participants will receive 1 injection of the IOP at Days 1,once time.
  Interventions: Drug: IOP Injection
- 0.9% normal saline (Placebo Comparator): Participants will receive 1 injection of 0.9% normal saline at Days 1,once time.
  Interventions: Drug: 0.9% normal saline

INTERVENTIONS:
Drug: IOP Injection — IOP Injection 20 mg Fe/ml, intravenous injection
  Other Names: Iron oxide nano particle m-PEG-silane
  Arms: IOP Injection
Drug: 0.9% normal saline — 0.9% normal saline 10 ml, intravenous injection
  Other Names: Sodium Chloride
  Arms: 0.9% normal saline

SUMMARY:
Study Objectives Primary: To determine MTD and dose limiting toxicities (DLTs) of IOP magnetic resonance imaging (MRI) contrast agent in healthy subjects.

Secondary:

1. To characterize the pharmacokinetic profiles of IOP MRI contrast agent in healthy subjects.
2. To evaluate safety/tolerability profiles of IOP MRI contrast agent in healthy subjects.
3. To explore efficacy profiles of IOP MRI contrast agent for liver organ in healthy subjects.

DETAILED DESCRIPTION:
Iron Oxide Nano Particle m-PEG-silane (IOP) Injection belongs to Superparamagnetic iron oxide (SPIO) can shorten the T2 relaxation time very effectively and reduces signal intensity in normal tissues. The mechanism of action increases after the particles have been phagocytosed by cells of the RES. Tissues with decreased RES function (e.g., metastases, primary liver cancer, cysts and various benign tumors, adenomas, and hyperplasia) retain their native signal intensity. In this study, investigators will characterize the PK profile, iron metabolism and preliminary efficacy of IOP Injection.

ELIGIBILITY:
Inclusion Criteria:

1. Male, age ≥ 20 ~40 years old with BMI between 18 and 27.
2. Subject must be in good general health condition (i.e., full physical examinations, medical history, vital signs, ECG, and clinical laboratory tests performed at screening) as determined by the investigator. Normal ECG is defined as normal cardiac conduction parameters including resting heart rate between 50 and 100 bpm, Fridericia-corrected QT interval (QTcF) ≤ 450 milliseconds, and QRS interval < 120 milliseconds.
3. Subject shows normal biochemistry test results (within normal range or considered clinically normal by the clinical investigator) at screening including items as listed below:

   * Blood urea nitrogen (BUN), creatinine, and uric acid.
   * Albumin and total protein.
   * Alkaline phosphatase, ALT,AST, and total bilirubin.
   * Serum iron, total iron-binding capacity, serum ferritin,percent transferrin saturation (TSAT), and transferrin.
   * Human immunodeficiency virus (HIV), Hepatitis B surface antigen (HBsAg), Antibody HBsAg (anti-HBs),and antibodies against HCV (anti-HCV).
4. Subject shows normal complete blood count (CBC) test results (within normal range or considered clinically normal by the clinical investigator) at screening including items as listed below:

   * Red blood cell (RBC) count and reticulocyte count.
   * White blood cell (WBC) count with differential.
   * Hemoglobin and hematocrit.
   * Platelet count.
5. Subject shows normal urinalysis test results (within normal range or considered clinically normal by the clinical investigator) at screening including items as listed below:

   * pH, color, appearance, and gravity
   * Erythrocyte, leukocyte, glucose, protein, ketones, and nitrite
   * Drug and alcohol abuse screening test including morphine, 3,4 methylenedioxymethamphetamine(MDMA), 3,4-methylenedioxyamphetamine (MDA),ketamine, codeine and alcohol.
6. Subject shows normal bleeding time test results (within normal range or considered clinically normal by the clinical investigator) at screening including prothrombin (PT) and activated partial thromboplastin time (APTT).
7. Male subjects must take reliable contraceptive method(s) during and after the study for a period of 14 days.
8. No screening of drug or alcohol abuse within one year prior to study enrollment.
9. Subjects are willing to comply with the protocol and sign informed consent form.

Exclusion Criteria:

1. Subjects have serious allergic history or known allergy to similar ingredients of the study contrast agent (i.e.,Gd-based and SPIO particles contrast agents).
2. Subjects have been diagnosed of Hepatitis B or C, venereal disease laboratory screens or have been determined of positive result of human immunodeficiency virus test.
3. Imaging and/or functional abnormalities of liver and/or spleen. That is,

   * Subjects have been diagnosed of abnormal liver function and appearances through medical histories, clinical laboratory tests, and imaging test including mild fatty liver, iron deposition or any acute/chronic liver change.
   * Subjects have signs of splenomegaly, enlargement of the spleen, or clinical laboratory tests showing signs of spleen functional abnormalities.
4. Subjects have been performed with any examinations with contrast agents applied within 28 days before study.
5. Subjects have alcohol or caffeine consumption within 48 hours prior to the administration of study contrast agent.
6. Subjects are unable to undergo an MRI scan.
7. Subjects have electronically, magnetically and mechanically activated implanted devices, including but not limited to automatic cardioverter defibrillators, cardiac pacemakers,insulin pumps, metallic splinters in the eye, ferromagnetic haemostatic clips in central nervous systems or vascular vessels.
8. Subjects have participated in other investigational trials within 28 days prior to study enrollment.
9. Subjects with active systemic infections, active and clinically significant cardiac diseases, active gastrointestinal ulcers, or medical conditions that may significantly affect action,adequate absorption and elimination of investigational contrast agent.
10. Subjects have taken any food 6 hours prior to administration.
11. Subject with conditions judged by the investigator as unsuitable for the study.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-02; Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLTs) of IOP | Up to 14 days post-IOP injection
  DLT is defined as any grade 2 or above toxicity by NCI-CTCAE version 4.03, as determined by the investigator and sponsor, to be at least possibly related in causality to the administered investigational product IOP
Maximum tolerated dose (MTD) of IOP | Up to 14 days post-IOP injection
  MTD is defined as the prior dose level below the dose level at which 2/6 subjects suffer dose limiting toxicities

SECONDARY OUTCOMES:
Pharmacokinetic parameters-Cmax | Up to 3 days post-IOP injection
  Cmax: the observed maximum drug concentration in plasma after dosing
Pharmacokinetic parameters-Tmax | Up to 3 days post-IOP injection
  Tmax: the time at which Cmax was reached
Pharmacokinetic parameters-AUC0-t | Up to 3 days post-IOP injection
  the truncated area under the plasma concentration-time curve from the beginning of dosing to time t
Pharmacokinetic parameters-AUC0-inf | Up to 3 days post-IOP injection
  the area under the plasma concentration-time curve from the beginning of dosing to time t (AUC0-t) extrapolated to time infinity
Pharmacokinetic parameters-T1/2 | Up to 3 days post-IOP injection
  terminal elimination half-life
Changes in laboratory safety tests (hematology, biochemistry, urinalysis, bleeding time) from baseline | Up to 14 days post-IOP injection

CONTACTS AND LOCATIONS:
Overall Officials: Rheun-Chuan Lee, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided